CLINICAL TRIAL: NCT02708537
Title: Effect of Plasma Rich in Growth Factors (PRGF) on Semen Quality
Brief Title: Effect of Plasma Rich in Growth Factors on Semen Quality
Status: Completed | Type: Observational
Sponsor: IVI Bilbao (Other)
Collaborators: bTI Vitoria (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1411-BIO-081-MF
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Vascular Endothelial Growth Factor Overexpression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PRGF in candidates for sperm donors: Prospective study of 58 candidates for sperm donors clinic IVI Bilbao.
  Interventions: Biological: PRGF in candidates for sperm donors

INTERVENTIONS:
Biological: PRGF in candidates for sperm donors — PRGF application on seminal aliquots will be conducted at different concentrations assessing sperm motility.

SUMMARY:
The hypothesis is growing semen samples with plasma rich in growth factors (PRGF), because it could improve sperm motility in patients subsidiary TRA, ultimately improving pregnancy rates.

DETAILED DESCRIPTION:
Platelet growth factors are a group of proteins involved in cellular communication modifying biological responses. Obtaining plasma rich in growth factors is already widespread and simple protocol technique that is being used in various areas of medicine with superb results. Described many of the growth factors present in the PRGF are related to sperm parameters, especially motility The described effects have been studied in mammalian and each growth factor individually. PRGF contains a pool of growth factors and therefore be interesting to analyze their effect on various sperm parameters.

One of those parameters is very important for fertilization sperm motility, since the lack of it will prevent displacement by the cervix to meet the egg in the fallopian tube.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years
* more than 5 million sperm per milliliter

Exclusion Criteria:

* Not having genetic and infectious diseases
* Do not suffer mental illness
* Have a family study determined that there is no risk of hereditary diseases
* There have fathered more than 6 children in the country

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prospective study of 58 candidates for sperm donors clinic IVI Bilbao.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the percentage of motile sperm adding PRGF versus those samples that growth factors were not added | 6 months
  Within concerted donor visits in IVI Bilbao will be held:
  * Removing Blood 9 mL of blood to obtain plasma rich in factors growth
  * Seminogram to analyze all semen parameters according to the criteria of the WHO (2010), paying particular attention to sperm motility.
  * Sperm vitality will be analyzed before and after treatment with PRGF. PRGF application on the seminal aliquots will be conducted at different concentrations assessing sperm motility.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Ferrando, Study Director — IVI Bilbao
Locations (2):
- Spain (2):
  - IVI Bilbao, Leioa, Vizcaya
  - BTI, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Yes
share data to BTI